CLINICAL TRIAL: NCT05209399
Title: Comparison of Ultrasound-guided Intraarticular Hip Injections With and Without Prior Local Anesthesia: a Randomized Controlled Trial
Brief Title: Comparison of Ultrasound-guided Intraarticular Hip Injections With and Without Prior Local Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: American Medical Society for Sports Medicine (Unknown)
Responsible Party: Principal Investigator, Rondy Lazaro, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00006887
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Hip Pain

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip injection with prior local anesthesia (Active Comparator)
  Interventions: Procedure: Ultrasound guided injection
- Hip injection without prior local anesthesia (Active Comparator)
  Interventions: Procedure: Ultrasound guided injection

INTERVENTIONS:
Procedure: Ultrasound guided injection — All intraarticular hip injections will be performed under real-time ultrasound guidance using a GE LOGIQ P9 ultrasound machine with a C1-5-RS 1-5 MHz curvilinear transducer (GE Healthcare, Chicago, IL, USA). For the procedure, patients will be placed in a supine position. The curvilinear transducer and ultrasound machine will be used to visualize the anterior aspect of the hip joint in a sagittal oblique plane. Sterile technique will be used to perform the procedure.

SUMMARY:
In this single-center randomized controlled trial, subjects undergoing a first-time ultrasound-guided unilateral intraarticular hip injection will be randomized into one of two groups: hip injection with prior local anesthesia (With LA) or hip injection without prior local anesthesia (Without LA). Visual analog scale (VAS) pain scores (0-100) will be collected after the local anesthesia injection (With LA group) and intraarticular hip injection (both groups). The primary outcome measure for comparison between the two groups will be VAS score for the intraarticular hip injection.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing a first-time ultrasound-guided unilateral intraarticular hip injection
* Subjects must be fluent in English
* Subject must be able to consent for themselves and mark pain levels on a visual analog scale.

Exclusion Criteria:

* previous intraarticular hip injection (to remove bias from prior injection experiences)
* prior surgery on the hip to be injected
* use of opioid medication on the day of or day before the procedure
* diabetes mellitus
* body mass index (BMI) greater than 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
mean pain score | baseline
  A visual analog pain score will be collected. The scale of the score is 0-100 with 100 indicating more pain.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center Physical Medicine and Rehabilitation, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lazaro RM, Smith JM, Bender N, Punreddy A, Barford N, Paul JH. Comparison of Pain With Ultrasound-Guided Intra-Articular Hip Injections With and Without Prior Subcutaneous Local Anesthesia. Clin J Sport Med. 2024 Jul 24;35(5):543-548. doi: 10.1097/JSM.0000000000001260. PMID 39046314